CLINICAL TRIAL: NCT02400112
Title: Local Application of Vancomycin Powder in Grade I-IIIA Open Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment; Low clinical relevance: evidence for use of vancomycin powder
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-111
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Fractures, Open; Surgical Wound Infection
Keywords: Vancomycin
MeSH Terms: conditions — Fractures, Open; Surgical Wound Infection | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin Powder (Experimental): If the patient randomizes to the experimental group (vancomycin powder), the patient will receive open fracture care identical to the control group except that, prior to closure, 1 gram of vancomycin powder will be applied locally to the open fracture bed. The traumatic and surgical wounds will be closed over a sterile drain and dressed, and the extremity will be immobilized.
  Interventions: Drug: Vancomycin
- Standard Treatment (No Intervention): If the patient randomizes to the control group (standard treatment), the patient will receive irrigation and debridement of the fracture site and surrounding soft tissues. The fracture will then be stabilized in standard fashion determined by fracture personality. Once stabilized, a sterile drain will be placed in the open fracture bed and the traumatic and surgical wounds will be closed and dressed. The extremity will then be immobilized.

INTERVENTIONS:
Drug: Vancomycin — Vancomycin powder administered locally, intraoperatively at site of open fracture
  Arms: Vancomycin Powder

SUMMARY:
The purpose of this study is to determine if local administration of vancomycin powder at the site of Grade I-IIIA open fractures at the time of surgery will be an efficacious method to lower infection rates in open fracture treatment and to elucidate any detrimental effects of applying vancomycin powder at the site of open fractures.

DETAILED DESCRIPTION:
Hypothesis:

Local administration of 1 gram of vancomycin powder at the site of primarily closeable Gustilo-Anderson Grade I-IIIA open fractures at the time of surgery, in addition to clinically accepted open fracture management (intravenous antibiotics, surgical irrigation and debridement and stabilization), will significantly decrease the postoperative infection rate in comparison to the current treatment algorithm.

Methods:

Study subjects will be randomized to one of two groups prior to surgery (parallel group design): standard treatment (control group) versus vancomycin powder treatment (experimental group). Each group will have an equal number of subjects. Once randomized, the intervention is then un-blinded to facilitate treatment.

Post-operatively, all patients will receive intravenous antibiotics, such that all patients receive a total of 24 hours of intravenous antibiotics. The surgical drain will be removed at the patient's bedside approximately 24 hours after the surgical procedure. Patients will follow up with their surgeon for routine scheduled visits at approximately 2 weeks, 6 weeks, 12 weeks, and further until aseptic union or resolution of infection. There will be no additional appointments solely for the purpose of research follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients ≥18 years of age
* Acute Gustilo-Anderson Type I-IIIA open fracture
* Fracture is deemed primarily closable at initial surgery
* Likely to follow-up with surgeon until fracture is healed
* Ability to understand and agree to Informed Consent

Exclusion Criteria:

* Patients <18 years of age
* Gustilo-Anderson Type IIIB and IIIC open fractures
* Open fractures requiring multiple operations (i.e. for repeat surgical debridement or staged bone grafting of critical segmental defects)
* Delayed presentation of open fracture
* Pre-existing systemic infection requiring antibiotic therapy
* Allergy to Vancomycin
* Open fracture at the site of a previous fracture or surgical site
* Current skin infection, chronic wounds or known systemic infection
* Unlikely to follow-up until fracture is healed
* Unable to understand or agree to Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Infection | one year
  Infections will be considered clinically significant if they require a return to the operating suite for surgical debridement. These infections will be classified as acute infections and/or chronic osteomyelitis. Superficial skin infections will be treated with local wound care, oral antibiotics and incision and drainage (as indicated). Deep infections and chronic osteomyelitis will be treated with staged serial surgical debridement, hardware removal (as indicated), culture specific IV antibiotics, and Infectious Disease consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk W Kiner, MD, Principal Investigator — University of Tennessee College of Medicine Chattanooga/Erlanger Health System
Locations (1):
- Erlanger Health System, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No